CLINICAL TRIAL: NCT05756335
Title: Quantifying the Brain Metabolism Underlying Task-Based BOLD Imaging
Brief Title: The Brain Metabolism of Unpredictable Signals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christin Y. Sander, PhD, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022P002851
Record Dates: First submitted 2023-02-15; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Brain metabolism; Positron Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral intervention (Experimental): Subjects are presented with a simultaneous sequence of faces and spoken words. Face stimuli include a representative sample of realistic faces across a range of ages. Spoken word stimuli are simple nouns spoken by a single female speaker.
  Interventions: Behavioral: (Un)predictable and (un)attended stimuli

INTERVENTIONS:
Behavioral: (Un)predictable and (un)attended stimuli — Subjects will complete four task conditions in each scan session: (1) Visual Unpredictable, (2) Visual Predictable, (3) Auditory Unpredictable, and (4) Auditory Predictable. In visual and auditory conditions subjects attend to visual or auditory stimuli and ignore the other domain, pressing a button when they detect an infrequently occurring stimulus inversion in the target domain. In unpredictable and predictable conditions, the attended domain either presents random (unpredictable) stimuli, or the same face or word stimuli repeated (predictable).

SUMMARY:
The investigators will be studying brain glucose and oxygen metabolism using hybrid PET/fMRI imaging to better understand how decoupling between brain glucose and oxygen metabolism relates to the processing of unpredictable sensory signals.

DETAILED DESCRIPTION:
The proposed research consists of one experiment, combining positron emission tomography (PET) and magnetic resonance imaging (MRI) techniques to simultaneously estimate the cerebral metabolic rates of glucose (CMRglc) and oxygen (CMRO2), and their ratio (oxygen:glucose index; OGI). These outcome measures will be collected in the context of a behavioral intervention presenting subjects with predictable and unpredictable stimuli, and attended and unattended stimuli. Functional PET uses a slow infusion of 2-[18F]-fluro-deoxyglucose (FDG) to estimate regional CMRglc, measuring relative changes in radiotracer uptake between blocks of task and rest. Dual-calibrated fMRI uses a sequence of hyperoxic (increased O2) and hypercapnic (increased CO2) challenges, along with a specialized sequence of MRI scans (estimating cerebral blood flow and blood-oxygen level-dependent signal) to estimate absolute CMRO2.

All subjects will be scanned, and each will complete the same behavioral intervention. First, the investigators will aim to assess the reliability of this hybrid imaging technique by having subjects complete two identical scan sessions. Second, the investigators will deliver a behavioral intervention to test the relationship between stimuli predictability, CMRglc, CMRO2, and OGI.

This experimental design is capable of producing effects observable in single subjects, and prior studies using fPET and dual-calibrated fMRI have produced effect sizes that our sample size is more than adequate to detect.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21-35.
* No contraindications to MRI or PET scanning.
* Right-handed.
* Fluent to speak, read, and understand English.

Exclusion Criteria:

* Adults unable to consent
* Contraindications to fMRI scanning and PET scanning (including the presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia)
* Inability to lie motionless in the scanner
* Pregnancy, seeking or suspecting pregnancy, or breastfeeding
* History of major head trauma
* Intracranial lesion
* Cardiovascular disorders, including heart disorders or high blood pressure [>155/95]
* Breathing problems such as severe asthma, emphysema, or pulmonary disease
* Bleeding disorder, or use of anticoagulants
* Bladder obstruction, urinary problems, or history of impaired elimination
* Known kidney or liver problems
* Past severe COVID-19 infection
* Intestinal blockage
* Raynaud syndrome
* Anemia
* Peripheral nerve injury
* Diabetes
* Glaucoma
* Current or recent use of medications (neurological or psychiatric) affecting brain function
* Current or past history of major medical, neurological, or psychiatric condition
* Current or past history of chronic pain (assessed at the discretion of PI)
* Current smoker
* Body mass index above 35
* Research-related radiation exposure exceeds current Radiology Department guidelines
* Lack of current health insurance coverage
* Employed under the direct supervision of the investigators conducting the research
* Unwilling or unable to cooperate with breathing maneuvers required during the gas challenge
* Respiratory or cardiac limitations to breathing at 20 L/min

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Brain positron emission tomography (PET) imaging signals | after PET image analysis and with study completion, an average of 1 year
  Changes in glucose metabolism will be quantified from brain PET images
Functional magnetic resonance imaging (fMRI) signals | after fMRI image analysis and with study completion, an average of 1 year
  Changes in oxygen metabolism will be quantified from dual-calibrated fMRI
Oxygen-glucose index | after PET/fMRI image analysis and with study completion, an average of 1 year
  Ratio of cerebral metabolic rates of glucose and oxygen from PET and fMRI signals

CONTACTS AND LOCATIONS:
Overall Officials: Christin Y Sander, PhD, Principal Investigator — Athinoula A. Martinos Center for Biomedical Imaging
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No